CLINICAL TRIAL: NCT02414009
Title: Open-label, Randomized, Multicenter, Phase II Trial to Compare Efficacy of CAPTEM Versus FOLFIRI as Second Line in Patients Progressed on or After First-line Oxaliplatin Chemo for Advanced, MGMT Methylated, RAS Mutated Colorectal Cancer
Brief Title: Study to Compare CAPTEM vs FOLFIRI as Second Line Treatment in Advanced, Colorectal Cancer Patients
Acronym: CAPTEM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAPTEM
Record Dates: First submitted 2015-02-05; First posted 2015-04-10 (Estimated); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine; Temozolomide; Irinotecan; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CAPTEM (Experimental): Patients in Arm A will receive capecitabine at the oral dose of 1500 mg/mq/die bid from day 1 to day 14 every 28 days plus temozolomide 150 mg/mq/die bid starting on day 10 to 14 every 28 days. Treatment will continue for up to 6 cycles or up to disease progression, unacceptable toxicity or informed consent withdrawal.
  Interventions: Drug: Capecitabine; Drug: Temozolomide
- FOLFIRI (Active Comparator): Patients in Arm B will receive FOLFIRI chemotherapy starting Day
  1 q2w (every cycle) starting on Day 1 of Cycle 1. FOLFIRI consists of irinotecan (starting dose of 180 mg/m2) on day one only; 5-FU 7 (starting bolus and 22-hour infusional doses of 400 mg/m2 and 600 mg/m2, respectively), and leucovorin (racemic, starting dose of 200 mg/m2 or L-form, starting dose of 100 mg/m2) for two consecutive days. Treatment will continue for up to 12 cycles in Arm B or up to disease progression, unacceptable toxicity or informed consent withdrawal.
  Interventions: Drug: Irinotecan; Drug: Fluorouracil; Drug: Leucovorin

INTERVENTIONS:
Drug: Capecitabine — Patients in Arm A will receive capecitabine at the oral dose of 1500 mg/mq/die refracted in two daily doses from day 1 to day 14 every 28 days
  Arms: CAPTEM
Drug: Temozolomide — Patients in Arm A will receive temozolomide 150 mg/mq/die refracted in two daily doses starting on day 10 to 14 every 28 days.
  Arms: CAPTEM
Drug: Irinotecan — Patients in Arm B will receive FOLFIRI chemotherapy starting Day 1 q2w (every cycle) starting on Day 1 of Cycle 1. FOLFIRI consists of irinotecan (starting dose of 180 mg/m2) on day one only; 5-FU (starting bolus and 22-hour infusional doses of 400 mg/m2 and 600 mg/m2, respectively), and leucovorin (racemic, starting dose of 200 mg/m2 or L-form, starting dose of 100 mg/m2) for two consecutive days.
  Arms: FOLFIRI
Drug: Fluorouracil — Patients in Arm B will receive FOLFIRI chemotherapy starting Day 1 q2w (every cycle) starting on Day 1 of Cycle 1. FOLFIRI consists of irinotecan (starting dose of 180 mg/m2) on day one only; 5-FU (starting bolus and 22-hour infusional doses of 400 mg/m2 and 600 mg/m2, respectively), and leucovorin (racemic, starting dose of 200 mg/m2 or L-form, starting dose of 100 mg/m2) for two consecutive days.
  Arms: FOLFIRI
Drug: Leucovorin — Patients in Arm B will receive FOLFIRI chemotherapy starting Day 1 q2w (every cycle) starting on Day 1 of Cycle 1. FOLFIRI consists of irinotecan (starting dose of 180 mg/m2) on day one only; 5-FU (starting bolus and 22-hour infusional doses of 400 mg/m2 and 600 mg/m2, respectively), and leucovorin (racemic, starting dose of 200 mg/m2 or L-form, starting dose of 100 mg/m2) for two consecutive days.
  Arms: FOLFIRI

SUMMARY:
Open-label, randomized, multicenter, Phase II trial designed to estimate the efficacy of CAPTEM versus FOLFIRI as second line treatment in MGMT methylated, RAS mutated advanced CRC patients who have progressed on or after first-line oxaliplatin containing chemotherapy for metastatic disease. MGMT will be assessed centrally at Pathology Department of Fondazione IRCCS Istituto Nazionale dei Tumori prior to enrollment. A minimum of ten 3-micron unstained sections on charged slides of tumor will be required and methylation status will be provided within a maximum of seven days to the Study Centers. Presence of RAS mutation will be assessed at each local participating center. Eligible patients will be randomized in a 1:1 ratio to one of two treatment arms:

* Arm A (experimental arm): CAPTEM
* Arm B (control arm): FOLFIRI Study treatment will be given in cycles repeated every 28 days for Arm A and every 14 days for Arm B. Patients in Arm A will receive capecitabine at the oral dose of 1500 mg/mq/die bid from day 1 to day 14 every 28 days plus temozolomide 150 mg/mq/die bid starting on day 9 to 14 every 28 days. Patients in Arm B will receive FOLFIRI chemotherapy starting Day 1 q2w (every cycle) starting on Day 1 of Cycle 1. FOLFIRI consists of irinotecan (starting dose of 180 mg/m2) on day one only; 5-FU 7 (starting bolus and 22-hour infusional doses of 400 mg/m2 and 600 mg/m2, respectively), and leucovorin (racemic, starting dose of 200 mg/m2 or L-form, starting dose of 100 mg/m2) for two consecutive days. Treatment will continue for up to 6 cycles in Arm A and up to 12 cycles in Arm B or up to disease progression, unacceptable toxicity or informed consent withdrawal. Randomization will be stratified across the treatment arms by the following predefined stratification variables: disease progression within 9 months from the start of first-line oxaliplatin-containing chemotherapy (< vs. ≥9 months); prior bevacizumab in combination with oxaliplatin-based chemotherapy (yes vs. no). Efficacy assessments will be performed every 2 cycles in Arm A and every 4 cycles in Arm B until progression. The study is expected to enrol approximately 82 patients who meet the eligibility criteria.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the third most commonly diagnosed cancer in males and the second in females, with over 1.2 million new cancer cases and 608,700 deaths estimated to have occurred in 2008. Approximately 35% of CRC patients present a Stage IV metastatic disease at the time of diagnosis, and 20%-50% of Stage II or III disease will progress to Stage IV at some point during the course of disease. Stage IV CRC carries a dismal prognosis: the 5-year survival rate is <10%, and median survival time of patients given optimal supportive care without chemotherapy is approximately 5 months. Hypothesis/rationale In advanced CRC, the occurrence of chemo- refractory disease poses a major therapeutic challenge for presence of an adequate performance status to potentially receive further treatments, but absence of effective drugs which may be offered to patients with an evidence-based algorithm. Patients who progress after all approved treatments may be generally considered suitable for new investigational drugs or strategies. Thus, in the era of personalized medicine, tumor molecular profiling may lead to the identification of therapeutic targets or predictive biomarkers for pharmacological intervention. The DNA repair gene O6-methylguanine-DNA methyltransferase (MGMT) is responsible of the elimination of alkyl groups from the O6-position of guanine. If inactive, it may be involved in early steps of colorectal tumorigenesis through an increase of the mutational rate particularly, G-to-A point mutations of KRAS gene. Epigenetic silencing of MGMT during colorectal tumorigenesis is associated with hypermethylation of the CpG island in its promoter. This transcriptional gene silencing is responsible for diminished DNA-repair of O6-alkylguanine adducts, with the consequence of enhancing chemosensitivity to alkylating agents in particular dacarbazine and its oral prodrug temozolomide. In a previous phase II study, the investigators showed that temozolomide induced an objective response rate by RECIST criteria in 12% of heavily pretreated patients with advanced CRC and MGMT promoter 6 methylation. Treatment was well tolerated, and the only grade 4 toxicity was one thrombocytopenia episode (3%). The trial met its primary end point of acceptable response rate, with a disease control rate of 31%, a median PFS (progression free survival) and OS (overall survival) of 1.8 and 8.4 months, respectively. Other studies in carcinoids cell lines demonstrated synergistic cell kill if 5-FU (5-fluorouracil) and TMZ (temozolomide) were delivered in a schedule-dependent manner. From these translational studies, it has been formulated the CAPTEM regimen using TMZ for 5 days at 150-200 mg/m2/day total daily dose on days 10-14 (given in BID oral dosing), with capecitabine 750 mg/m2 PO (per OS) BID on days 1-14 of a 28-day cycle. The use of TMZ in BID (BIS in DIE) dosing instead of daily dosing was done because the first dose binds 6-MGMT levels, thus allowing the second dose to methylate guanines with decreased repair from MGMT. Given the potential synergy of CAPTEM combination in CRC, the investigators planned a randomized study of second-line CAPTEM vs. FOLFIRI after failure of prior first-line oxaliplatin - based treatment. Study design Open-label, randomized, multicenter, Phase II trial designed to estimate the efficacy of CAPTEM versus FOLFIRI as second line treatment in MGMT methylated, RAS mutated advanced CRC patients who have progressed on or after first-line oxaliplatin containing chemotherapy for metastatic disease. MGMT will be assessed centrally at Pathology Department of Fondazione IRCCS Istituto Nazionale dei Tumori prior to enrollment. A minimum of ten 3-micron unstained sections on charged slides of tumor will be required and methylation status will be provided within a maximum of seven days to the Study Centers. Presence of RAS mutation will be assessed at each local participating center. Eligible patients will be randomized in a 1:1 ratio to one of two treatment arms:

* Arm A (experimental arm): CAPTEM
* Arm B (control arm): FOLFIRI Study treatment will be given in cycles repeated every 28 days for Arm A and every 14 days for Arm B. Patients in Arm A will receive capecitabine at the oral dose of 1500 mg/mq/die bid from day 1 to day 14 every 28 days plus temozolomide 150 mg/mq/die bid starting on day 10 to 14 every 28 days. Patients in Arm B will receive FOLFIRI chemotherapy starting Day

  1 q2w (every cycle) starting on Day 1 of Cycle 1. FOLFIRI consists of irinotecan (starting dose of 180 mg/m2) on day one only; 5-FU 7 (starting bolus and 22-hour infusional doses of 400 mg/m2 and 600 mg/m2, respectively), and leucovorin (racemic, starting dose of 200 mg/m2 or L-form, starting dose of 100 mg/m2) for two consecutive days. Treatment will continue for up to 6 cycles in Arm A and up to 12 cycles in Arm B or up to disease progression, unacceptable toxicity or informed consent withdrawal. Randomization will be stratified across the treatment arms by the following predefined stratification variables: disease progression within 9 months from the start of first-line oxaliplatin-containing chemotherapy (< vs. ≥9 months); prior bevacizumab in combination with oxaliplatin-based chemotherapy (yes vs. no). Efficacy assessments will be performed every 2 cycles in Arm A and every 4 cycles in Arm B until progression. The study is expected to enrol approximately 82 patients who meet the eligibility criteria. Number of study centres 10 centers in Italy Primary objective and corresponding end point
* To evaluate the efficacy, as measured by progression-free survival, of FOLFIRI (administered every 2 weeks) versus CAPTEM (administered four-weekly) Secondary objectives and corresponding end points
* To evaluate the activity of the two regimens, as measured by response rate; secondary efficacy endpoints also include duration of response and overall survival of FOLFIRI (administered every 2 weeks) versus CAPTEM (administered four-weekly)
* To evaluate the safety of FOLFIRI versus CAPTEM
* To assess the quality of life as measured by Quality of life questionnaires (EORTC QLQ - CR29; QLQ-C30) Statistical methodology According to the published results of the GERCOR study, the median progression-free survival during second-line treatment with crossover from FOLFOX to FOLFIRI was 2.3 months (calculated from the start of second-line treatment with FOLFIRI). A one-sided log rank test with an overall sample size of 82 subjects (41 in the control group and 41 in the study group) achieves 90% power at a 5% significance level to detect an increase in median progression free survival from 2 months of the control group to 4 months. The study lasts for 30 months of which subject accrual (entry) occurs in 24 months

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Histologically or cytologically confirmed adenocarcinoma of the colon and/or rectum, with MGMT promoter methylation and RAS mutation.
* Progressive disease on or after a first-line oxaliplatin containing chemotherapy regimen for mCRC with or without bevacizumab or other anti-angiogenic drugs. Patients must have received oxaliplatin-containing chemotherapy for ≥ 3 months. No more than one prior chemotherapy regimen for metastatic disease is allowed. 8
* Disease measurableRECIST v1.1
* Age ≥ 18 years and ≤ 75 years
* Life expectancy ≥ 12 weeks
* ECOG Performance Status of 0 1
* Adequate hematologic and end-organ function, defined by laboratory results obtained within 14 days prior to first administration: ANC ≥ 1500/μL Platelet count ≥ 100,000/μL Hemoglobin ≥ 9.0 g/dL Albumin ≥ 2.5 g/dL
* Total bilirubin ≤ 1.5 × the upper limit of normal (ULN)
* AST, ALT, and/or alkaline phosphatase ≤ 2.5 × ULN, with the following exceptions: Patients with documented hepatic metastases are eligible with AST, ALT, and/or alkaline phosphatase ≤ 5 × ULN. Patients with documented bone metastases are eligible with alkaline phosphatase ≤ 5 × ULN.
* Serum creatinine ≤ 1.5 × ULN, or creatinine clearance ≥ 50 mL/min on the basis of the Cockcroft-Gault glomerular filtration rate estimation: (140 - age) × (weight in kg) × (0.85 if female) 72 × (serum creatinine in mg/dL)
* INR and aPTT ≤ 1.5 × ULN
* documented agreement (by patient and/or partner) to use an effective means of contraception (e.g., surgical sterilization, a reliable barrier method, birth control pills, or contraceptive hormone implants) and to continue its use for the duration of the study and for 60 days for female patients or 150 days for male patients with partners of childbearing potential after the last infusion of study treatment.
* Consent to provide mandatory archival tumor tissue for biomarker testing

Exclusion Criteria:

* Prior treatment with irinotecan and temozolomide
* Major surgical procedure within 4 weeks and radiotherapy within 2 weeks prior to Day 1 Cycle 1
* Symptomatic hypercalcemia requiring continued use of bisphosphonate.
* Known clinically significant dihydropyrimidine 9 dehydrogenase deficiency
* Current severe, uncontrolled systemic disease Active infection requiring IV antibiotics
* History of heart failure of any New York Heart Association criteria or serious cardiac arrhythmia requiring treatment (except for atrial fibrillation and paroxysmal supraventricular tachycardia)
* History of myocardial infarction within 6 months prior to Cycle 1, Day 1, or history of unstable angina
* Known clinically significant liver disease,or current alcohol abuse
* History of bleeding diathesis or coagulopathy other than that due to anticoagulation therapy
* Patients receiving oral coumarin-derived anticoagulants
* Active haemoptysis within 30 days prior to Cycle 1, Day 1
* HIV infection
* Untreated/active CNS metastases (progressing or requiring anticonvulsants or corticosteroids for symptomatic control). Patients with a history of treated CNS metastases are eligible provided they meet all of the following criteria: Measurable disease outside the CNS as defined by RECIST v1.1.Radiotherapy completed ≥ 4 weeks prior to Cycle, 1 Day
* Pregnancy or lactation. Women of childbearing potential (including those who have had a tubal ligation) must have a documented negative serum pregnancy test within 14 days prior to Cycle 1, Day 1.
* Inability to take oral medications.
* Malignancies other than CRC within 3 years prior to randomization, with the exception of adequately treated basal or squamous cell skin cancer and carcinoma in situ of the cervix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2014-09; Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Progression-free survival of FOLFIRI versus CAPTEM | 30 months
  evaluate the efficacy, measured by progression-free survival, of FOLFIRI (administered every 2 weeks) versus CAPTEM (administered four-weekly)

SECONDARY OUTCOMES:
Response rate | 30 months
  Evaluation of activity of the two regimens, as measured by response rate.
Overall survival of FOLFIRI versus CAPTEM | 30 months
  include duration of response and overall survival of FOLFIRI (administered every 2 weeks) versus CAPTEM (administered four-weekly)
Number of Adverse events | 30 months
  Assess adverse events by CTCAE version 4.0
Quality of life measured by QLQ-C30 | 30 months
  Assess the quality of life as measured by QLQ-C30
Quality of life measured by EORTC FACT-C | 30 months
  Assess the quality of life as measured by EORTC FACT-C

CONTACTS AND LOCATIONS:
Overall Officials: Filippo de Braud, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale Tumori, Milan, Mi, Italy